CLINICAL TRIAL: NCT02370836
Title: Evaluating the Effects of Psycho-oncological Education on Distress and Quality of Life in Solid Tumor Patients Who Have Received and Completed Chemotherapy Treatment With Curative Intent. A Pilot Study.
Brief Title: Evaluating the Effects of Psycho-oncological Education on Distress and Quality of Life in Solid Tumor Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SIB14142
Record Dates: First submitted 2015-02-03; First posted 2015-02-25 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Quality of Life
Keywords: distress
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psycho-oncological education (Experimental): One 60 minute psycho-oncological education session on late effects, fatigue and stress management.
  Interventions: Other: Education
- Usual Care (No Intervention): Usual care includes completion of a symptom checklist by the nurse practitioner

INTERVENTIONS:
Other: Education — One 60 minute psycho-oncological educational session on stress management, late effects and fatigue.
  Arms: Psycho-oncological education

SUMMARY:
This study evaluates that effects of psycho-oncological education on distress and quality of life in solid tumor cancer patients who have completed chemotherapy with curative intent. Half of the participants will received a psycho-oncological educational intervention while the other half will receive usual care.

DETAILED DESCRIPTION:
Solid tumor cancer patients who have completed chemotherapy with curative intent experience psychological distress. As a result these patients experience poorer quality of life (QOL), emotional vulnerability and unnecessary emotional suffering.

Purpose: To determine whether the implementation of a nurse driven psycho-oncological educational session will decrease psychological distress levels and improve QOL among solid tumor cancer patients who have received and completed chemotherapy with curative intent.

Methods: A randomized clinical trial (RCT) consisting of 28 eligible patients at Sibley Memorial Hospital will be used to compare the effect of psycho-oncological education to treatment as usual in reducing psychological distress and improving quality of life. The intervention group will receive one 60 minute session of psycho-oncological education. The comparison group will receive usual care only which includes a general information session offered prior to any treatment which addresses broad side-effects of treatment, an overview of the treatment process and identification of additional resources. Participants will be assessed for psychological distress and QOL levels at baseline and two weeks after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* non-race specific
* solid tumor cancer patient
* completed chemotherapy with curative intent

Exclusion Criteria:

* diagnosis of cancer prior to cancer they are being treated for
* distress score of 8 or greater
* diagnosed with a psychiatric disorder
* diagnosed with lymphoma or leukemia
* in need of immediate crisis support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Distress Thermometer (self-reported distress levels by 11 point scale) Change is being assessed | at baseline & two weeks after intervention
  Self reported distress levels at baseline and two weeks after the intervention. Scale is 11-points from 0(no distress) to 10 (extreme distress)

SECONDARY OUTCOMES:
World Health Organization Quality of Life BREF (WHOQOL-BREF) Change is being assessed. | at baseline & two weeks after intervention
  Self- report, 24 question scale representing 6 domains related to quality of life. Quality of life to be measured at baseline and two weeks post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Channing Paller, MD, Principal Investigator — Johns Hopkins University